CLINICAL TRIAL: NCT06471543
Title: A Phase 1, Randomized, Placebo-controlled, Single Ascending Dose and Phase 2 Randomized, Placebo Controlled, Parallel-Group, Single-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamic Effects, and Immunogenicity of RN0361 in Adult Healthy Subjects and Hypertriglyceridemic Subjects
Brief Title: Study of RN0361in Adult Healthy Subjects and Adult Hypertriglyceridemic Subjects
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ikaria Bioscience Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RN0361-101
Record Dates: First submitted 2024-06-06; First posted 2024-06-24 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hypertriglyceridemia; Familial Chylomicronemia Syndrome
MeSH Terms: conditions — Hypertriglyceridemia; Familial hyperchylomicronemia syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RN0361 (Experimental): subcutaneous injections
  Interventions: Drug: RN0361
- Placebo (Placebo Comparator): calculated volume to match active treatment
  Interventions: Drug: RN0361

INTERVENTIONS:
Drug: RN0361 — Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and immunogenicity of single doses of RN0361 in Adult healthy subjects and Adult Hypertriglyceridemic Subjects.

ELIGIBILITY:
Phase I：

Inclusion Criteria:

* Willing to provide written informed consent before any study-specific procedures.
* Comply with the study requirements and restrictions as listed in the Informed Consent Form and the protocol.
* Fasting serum triglyceride levels > 80 mg/dL and fasting LDL-C ≥70 mg/dL at screening
* Female participants must either be nonchildbearing or, if of childbearing potential, not pregnant, not breastfeeding, and using effective contraception. Male participants must use condoms and ensure their partners use contraception if they are of childbearing potential.
* Participants must avoid sperm or egg donation during the study

Exclusion Criteria:

* History or presence of any serious or uncontrolled disease
* clinically significant health concerns
* Recent vaccination with live vaccines, except for influenza, or plans to receive such during the study.
* Positive tests for alcohol or drugs of abuse at screening.
* History of multiple drug allergies or allergic reactions to specific components used in the study.

Phase II:

Inclusion Criteria:

* Willing to provide written informed consent before any study-specific procedures.
* Comply with the study requirements and restrictions as listed in the Informed Consent Form and the protocol.
* Fasting serum triglyceride levels ≥ 300 mg/dL at screening
* Female participants must either be nonchildbearing or, if of childbearing potential, not pregnant, not breastfeeding, and using effective contraception. Male participants must use condoms and ensure their partners use contraception if they are of childbearing potential.

Exclusion Criteria:

* History or presence of any serious or uncontrolled disease
* Active pancreatitis within 12 weeks prior to Day 1
* Uncontrolled hypertension (sitting blood pressure) >160/100 mm Hg
* Uncontrolled diabetes
* Symptomatic heart failure (NYHA II-IV)
* Positive serologic test of HBV, HCV, or HIV
* Alcohol or drugs abuse
* History of multiple drug allergies or history of allergic reaction to an oligonucleotide or GalNAc.
* History of intolerance to SC injection or relevant abdominal scarring (surgical, burns, etc)
* History of malignancy within the last 2 years prior to the date of consent

Note: Additional inclusion/exclusion ceiteria may apply, per protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-06-03 (Estimated); Study Completion 2026-08-26 (Estimated)

PRIMARY OUTCOMES:
Number and incidence of adverse events (AEs)/serious adverse events (SAEs) possibly or probably related to treatment of RN0361 in adult healthy subjects. | Up to Day85
  Phase 1
Absolute and percent change from baseline in APOC3 and fasting triglycerides (TG) in subjects with HTG | Up to Day183
  Phase 2

SECONDARY OUTCOMES:
Plasma pharmacokinetics (PK) parameters (Cmax) of a single ascending SC dose of RN0361 and its metabolite AS3'N-1 in adult healthy subjects. | Up to 48 hours post-dose
  Phase 1
Plasma pharmacokinetics (PK) parameters (Tmax) of a single ascending SC dose of RN0361 and its metabolite AS3'N-1 in adult healthy subjects. | Up to 48 hours post-dose
  Phase 1
Plasma pharmacokinetics (PK) parameters (AUC 0-24) of a single ascending SC dose of RN0361 and its metabolite AS3'N-1 in adult healthy subjects. | Up to 48 hours post-dose
  Phase 1
Plasma pharmacokinetics (PK) parameters (t1/2) of a single ascending SC dose of RN0361 and its metabolite AS3'N-1 in adult healthy subjects. | Up to 48 hours post-dose
  Phase 1
Plasma pharmacokinetics (PK) parameters (AUC0-inf) of a single ascending SC dose of RN0361 and its metabolite AS3'N-1 in adult healthy subjects. | Up to 48 hours post-dose
  Phase 1
Plasma pharmacokinetics (PK) parameters (Vz/F) of a single ascending SC dose of RN0361 and its metabolite AS3'N-1 in adult healthy subjects. | Up to 48 hours post-dose
  Phase 1
Plasma pharmacokinetics (PK) parameters (λz) of a single ascending SC dose of RN0361 and its metabolite AS3'N-1 in adult healthy subjects. | Up to 48 hours post-dose
  Phase 1
Urine pharmacokinetics (PK) parameters (CLR) of a single ascending SC dose of RN0361 and its metabolite AS3'N-1 in adult healthy subjects. | Up to Day 85
  Phase 1
Urine pharmacokinetics (PK) parameters (Aet) of a single ascending SC dose of RN0361 and its metabolite AS3'N-1 in adult healthy subjects. | Up to Day 85
  Phase 1
Urine pharmacokinetics (PK) parameters (Aeu) of a single ascending SC dose of RN0361 and its metabolite AS3'N-1 in adult healthy subjects. | Up to Day 85
  Phase 1
Urine pharmacokinetics (PK) parameters (FE) of a single ascending SC dose of RN0361 and its metabolite AS3'N-1 in adult healthy subjects. | Up to Day 85
  Phase 1
Absolute and percent change from baseline in APOC3 in adult healthy subjects. | Up to Day 85
  Phase 1
Absolute and percent change from baseline in TG in adult healthy subjects. | Up to Day 85
  Phase 1
Number and incidence of adverse events (AEs)/serious adverse events (SAEs) possibly or probably related to treatment of RN0361 in subjects with HTG. | Up to Day 183
  Phase 2
Absolute and percent change from baseline in remnant cholesterol and VLDL-C in subjects with HTG. | Up to Day 183
  Phase 2

CONTACTS AND LOCATIONS:
Locations (10):
- United States (6):
  - TBC Research LLC,, Tamarac, Florida
  - Versailles Family Medicine / Avacare, Versailles, Kentucky
  - Axis Clinicals USA, Dilworth, Minnesota
  - Synergy Groups Medical, Houston, Texas
  - Tranquil, Webster, Texas
  - Ogden Clinic, Mountain View / Avacare, Pleasant View, Utah
- Australia (4):
  - University of the Sunshine Coast Clinical Trials, Morayfield, Queensland
  - University of the Sunshine Coast Clinical Trials, Sippy Downs, Sippy Downs, Queensland
  - Altona Clinical Research, Altona N., Victoria
  - Nucleus Network Melbourne, Melbourne, Victoria